CLINICAL TRIAL: NCT01261585
Title: Study of the Modification of the Fixation of FDG, F-Miso and FLT Measured in PET/CT at Patients Before and in the Course of Exclusive Radiotherapy or Concomitant Radiochemotherapy for Primitive Bronchial Cancer
Brief Title: Study of the Fixation of Various Vectors in PET/CT in Patients With a With Lung Cancer Before and During of CRT or RT
Acronym: RTEP4
Status: Completed | Type: Observational
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Mohamed GUERNOU MD, Centre Henri Becquerel
Other Study IDs: CHB 08-01
Record Dates: First submitted 2010-12-15; First posted 2010-12-16 (Estimated); Last update posted 2010-12-16 (Estimated); Status verified 2009-01

CONDITIONS: Bronchial Neoplasms; Carcinoma, Non-Small-Cell Lung
Keywords: Positron-Emission Tomography; PET Scan; FDG; FLT; FMISO; Non-Small-Cell Lung Carcinoma; chemo-Radiation Oncology; SUV
MeSH Terms: conditions — Bronchial Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Study of the modification of the fixation(binding) of Fluoro-2-deoxy-D-glucose (FDG), fluoro-misonidazole (FMISO) and 3'deoxy-3-fluoro-thymidine deoxy-3-fluoro-thymidine (FLT) measured in tomography by broadcast(emission,issue) of positrons (PET) at patients before and in the course of exclusive radiotherapy or concomitant radiochemotherapy for primitive bronchial cancer.

This protocle allows to study the simultaneous variations of the metabolism, the hypoxie and the cellular proliferation by PET SCAN at 5 patients reached(affected) by a primitive bronchial cancer in the course of exclusive radiotherapy for primitive bronchial cancer not small cell lung.

The investigators are also going to study several scenarii of optimization of the radiotherapy according to the variations of the tumoral metabolism, the hypoxie and the cellular proliferation measured in the course of radiotherapy (theoretical study on console using the scanner and the various examinations).

ELIGIBILITY:
Inclusion Criteria:

* patients with non-small-cell lung carcinoma hitologicaly proved
* Candidate patients in a treatment with aim guardian by exclusive thoracic radiotherapy or of concomitant radiochemotherapy (tumoral dose superior to 60 Gy) ( n=5 ).
* Measurable tumor according to the criteria of evaluation RECIST

Exclusion Criteria:

* Histology other one than primitive bronchial cancer not in small cells lung
* The patients for whom no tumoral target is assessable (forgiveness completes after first chemotherapy, operated patients).
* Patients for whom a radiotherapy with curative aim is not indicated (tumoral extension, metastases, general state, co-morbidity).
* Patient having benefited from an examination PET in the FDG with in more than 4 weeks and for which a new PET in the FDG is not necessary with in the framework of its disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosed patients with non-small-cell lung carcinoma
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2008-12; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GUERNOU Mohamed, MD, Principal Investigator — CHBecquerel; VERA Pierre, MD phD, Study Director — CHBecquerel
Locations (1):
- Centre Henri Becquerel, Rouen, Hate Normandie, France

REFERENCES:
- [Derived] Ganem J, Thureau S, Gardin I, Modzelewski R, Hapdey S, Vera P. Delineation of lung cancer with FDG PET/CT during radiation therapy. Radiat Oncol. 2018 Nov 12;13(1):219. doi: 10.1186/s13014-018-1163-2. PMID 30419929
- [Derived] Calais J, Thureau S, Dubray B, Modzelewski R, Thiberville L, Gardin I, Vera P. Areas of high 18F-FDG uptake on preradiotherapy PET/CT identify preferential sites of local relapse after chemoradiotherapy for non-small cell lung cancer. J Nucl Med. 2015 Feb;56(2):196-203. doi: 10.2967/jnumed.114.144253. Epub 2015 Jan 8. PMID 25572091